CLINICAL TRIAL: NCT06538766
Title: Strength Training for Gait Rehabilitation in Older Adults: Insights From Neuroscience
Brief Title: The Effect of Different Focus of Attention Instructions on Resistance Training and Its Transfer to Gait Parameters in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1236- Fractal of attention
Record Dates: First submitted 2024-07-26; First posted 2024-08-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging; Healthy
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Internal Focus Condition (Active Comparator): In the internal focus condition the participant is instructed to realize seated calf raises by focusing on contracting the plantar-flexors. In clinical applications the internal focus is the most commonly used instruction. It is not possible to have a neutral focus condition, as participants always have to receive instructions and will always be focusing on something. Therefore, the internal focus condition is used as an active comparator.
  Interventions: Other: Strength training with an internal focus of attention
- Proprioceptive External Focus Condition (Experimental): In the proprioceptive external focus condition the participant is instructed to realize seated calf raises by focusing on lifting the machine's bar.
  Interventions: Other: Strength training with a proprioceptive external focus of attention
- Visual External Focus Condition (Experimental): In the visual external focus condition the participant is instructed to realize seated calf raises by focusing on a line representing the displacement of the bar projected on a screen.
  Interventions: Other: Strength training with a visual external focus of attention

INTERVENTIONS:
Other: Strength training with an internal focus of attention — A 4 weeks strength training program of seated calf raises with progressive overload is carried out. A supervisor applies force specific internal focus instruction in three sessions per week with at least 48h rest time. One session consists of 3 series until failure with 75%RM. Rest intervals between series are defined as 2 minutes.
  Arms: Internal Focus Condition
Other: Strength training with a proprioceptive external focus of attention — A 4 weeks strength training program of seated calf raises with progressive overload is carried out. A supervisor applies force specific proprioceptive external focus instruction in three sessions per week with at least 48h rest time. One session consists of 3 series until failure with 75%RM. Rest intervals between series are defined as 2 minutes.
  Arms: Proprioceptive External Focus Condition
Other: Strength training with a visual external focus of attention — A 4 weeks strength training program of seated calf raises with progressive overload is carried out. A supervisor applies force specific visual external focus instruction in three sessions per week with at least 48h rest time. One session consists of 3 series until failure with 75%RM. Rest intervals between series are defined as 2 minutes.
  Arms: Visual External Focus Condition

SUMMARY:
The goal of this clinical trial is to investigate the effects of strength training with different focus of attention strategies on plantar flexor force and how this affects gait in apparently healthy older adults. The main questions it aims to answer are:

* Is there an acute effect of focus of attention on non-linear force variability and the subjacent neurophysiological mechanisms in apparently healthy young and older adults?
* Is there a training effect of focus of attention on non-linear force variability and does it transfer to non-linear gait variability as well as the respective subjacent neurophysiological mechanisms in apparently healthy older adults?

Researchers will compare two different external focus strategies with an internal focus to see if non-linear variability increases and subjacent neurophysiological mechanisms are more automized with an external focus of attention compared to an internal focus. In the acute study young adults are assessed as the differences between focus conditions are thought to be in the same direction as for older adults but attenuated.

Participants will carry out training and strength assessments of the calf muscles and walking on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

- Signed informed consent

Exclusion Criteria:

* Severe cardiovascular or pulmonary disease
* Oncological disease
* Lower limb disabilities
* Neurological disorders
* Inability to walk unassisted for 12 continuous minutes
* Cognitive impairment
* Falls in the prior 12 months
* Orthopedic concerns, which might limit force production
* Metal implants
* Medicine that can trigger side effects with TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Non-linear Force Variability after each Week during Intervention and 2 Weeks Follow-Up | Baseline, Week1, Week2, Week3, Week4 and Follow-Up (Week6)
  The non-linear variability of the temporal structure of the force signal of a 50 seconds isometric task at 50% of the maximum voluntary isometric contraction is analyzed using sample entropy (SampEn), which indicates the probability that short sequences of data points are repeated throughout the signal length. Lower SampEn (towards 0) is the consequence of similar distances between repetitions of those sequences, which indicates a more regular force output. A higher SampEn value (towards infinity) results from large differences of distances between repetitions of sequences, which designates a more irregular, variable force output.
Change from Baseline in Non-linear Gait Variability after each Week during Intervention and 2 Weeks Follow-Up | Baseline, Week1, Week2, Week3, Week4 and Follow-Up (Week6)
  The non-linear variability of the temporal structure of the gait signal from a 12 minutes gait trial is analyzed using sample entropy (SampEn), which indicates the probability that short sequences of data points are repeated throughout the signal length. Lower SampEn (towards 0) is the consequence of similar distances between repetitions of those sequences, which indicates a more regular gait output. A higher SampEn value (towards infinity) results from large differences of distances between repetitions of sequences, which designates a more irregular, variable gait output.
Change from Baseline in Cortico-Spinal Excitability after 2 Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  The cortical measures are assessed with transcranial magnetic stimulation (TMS). A stimulator generates motor evoked potentials (MEP) in the active soleus muscle during a low-intensity plantarflexion. To assess cortico-spinal excitability single-pulse TMS is applied. For cortico-spinal excitability the mean of the MEP amplitude from 10 stimulations is calculated. The values will be presented in % normalized to the EMG maximum voluntary contraction.
Change from Baseline in Cortico-Spinal Inhibition after 2 Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  The cortical measures are assessed with transcranial magnetic stimulation (TMS). A stimulator generates motor evoked potentials (MEP) in the active soleus muscle during a low-intensity plantarflexion. To assess cortico-spinal inhibition single-pulse TMS is applied. For cortico-spinal inhibition the mean of electromyographic silent periods from 10 stimulations is calculated. The values are presented in ms.
Change from Baseline in Intra-Cortical Inhibition after 2 Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  The cortical measures are assessed with transcranial magnetic stimulation (TMS). A stimulator generates motor evoked potentials (MEP) in the active soleus muscle during a low-intensity plantarflexion. To assess intra-cortical inhibition paired-pulse TMS is applied. For intra-cortical inhibition the mean of the MEP amplitude from 10 stimulations is calculated. The values will be presented in % normalized to the cortico-spinal excitability.
Change from Baseline in Intra-Cortical Facilitation after 2 Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  The cortical measures are assessed with transcranial magnetic stimulation (TMS). A stimulator generates motor evoked potentials (MEP) in the active soleus muscle during a low-intensity plantarflexion. To assess intra-cortical facilitation paired-pulse TMS is applied. For intra-cortical facilitation the mean of the MEP amplitude from 10 stimulations is calculated. The values will be presented in % normalized to the cortico-spinal excitability.

SECONDARY OUTCOMES:
Change from Baseline in Antagonist Co-Contraction Index after 2Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  The antagonist co-contraction index (CCI) of the soleus as well as of the lateral and medial gastrocnemius heads with tibialis anterior will be calculated based on the formula: CCI=lowEMG/highEMG×(highEMG+lowEMG).
Change from Baseline in Linear Force Variability after each Week during Intervention and 2 Weeks Follow-Up | Baseline, Week1, Week2, Week3, Week4 and Follow-Up (Week6)
  The linear measure of variability is analyzed with the coefficient of variation (CV), which indicates the amount of variability within the force signal.
Change from Baseline in Linear Gait Variability after each Week during Intervention and 2 Weeks Follow-Up | Baseline, Week1, Week2, Week3, Week4 and Follow-Up (Week6)
  The linear measure of variability is analyzed with the coefficient of variation (CV), which indicates the amount of variability within the gait signal.
Change from Baseline of Hip, Knee, Ankle Range of Motion during Gait after 2Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  Hip, knee, ankle range of motion during gait will be assessed using a motion capture system. This analysis assesses the angular displacement of each joint through the different phases of the gait cycle. For the hip and knee joint the ROM involves flexion and extension, while for the ankle joint dorsiflexion and plantarflexion are measured.
Change from Baseline of Minimum Toe Clearance during Gait after after 2Weeks, 4 Weeks of Intervention and 2 Weeks Follow-Up | Baseline, Week2, Week4 and Follow-Up (Week6)
  Minimum toe clearance during gait will be assessed using a motion capture system. This analysis measures the smallest vertical distance between the toe and the ground during the swing phase of the gait cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health & Science, Monte de Caparica, Almada, Portugal